CLINICAL TRIAL: NCT04088669
Title: Efficiency of Home-Based Pulmonary Rehabilitation in Adults With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ayşe Sena Manzak, Research Asisstant, PhD, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BVUaysesena01
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Rehabilitation; Asthma; Home-based Pulmonary Rehabilitation
Keywords: asthma; pulmonary rehabilitation; home-based pulmonary rehabilitation; home-based rehabilitation
MeSH Terms: conditions — Asthma | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A home-based pulmonary rehabilitation program for 8 weeks, with a minimum of 3 days per week and one session of this is under the supervision of a physiotherapist.
  Interventions: Other: Home-based Pulmonary Rehabilitation
- Control group (Active Comparator): A training session about the disease and the correct inhaler use, booklets that include physical activity recommendations.
  Interventions: Other: Education and Recommendations

INTERVENTIONS:
Other: Home-based Pulmonary Rehabilitation — Patients will admit a home-based pulmonary rehabilitation program for 8 weeks, with a minimum of 3 days per week and one session of this is under the supervision of a physiotherapist. The pulmonary rehabilitation program includes stretching exercises, strengthening exercises for upper and lower extremities, breathing exercises and aerobic exercises (walking). All of these exercises will be equipped with equipment that the patients can easily provide at home. In addition, patients will be provided with a pedometer and exercise diary.
  Arms: Intervention group
Other: Education and Recommendations — The control group will be given a training session on the course of the disease and the correct inhaler use and will be given booklets on physical activity recommendations. Patients will be given a pedometer and diary.
  Arms: Control group

SUMMARY:
Asthma is a serious global health problem affecting people of all ages in every country in the world. Despite the presence of effective medications, many studies have reported poor asthma control in patients. Therefore, new approaches are needed to improve asthma control. Pulmonary rehabilitation is recommended as an alternative approach in patients with chronic lung disease including asthma. Also, home-based type of pulmonary rehabilitation can be preferred because it is more cost-effective and patients can spend more time with their families. There are a limited number of studies in the literature evaluating the efficacy of home-based pulmonary rehabilitation in asthmatic patients. The aim of this study was to investigate the efficacy of home-based pulmonary rehabilitation program with simple equipment in asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with asthma
* Acceptance of persons to participate in the study
* Being in the 18-65 age range

Exclusion Criteria:

* Presence of an orthopedic, neurological, systemic disease that prevents the exercise
* Having mental, communicative and behavioral disorders that may cause problems in understanding commands and questions or practicing exercises.
* Exercising 3 or more days a week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 8 weeks
  Change of Six-Minute Walking Test Distance from baseline to 8 weeks.The distance covered in meters in a straight corridor of 30 meters will be recorded as fast as possible but without running for 6 minutes. The distance that normal individuals should take in this period is 400-700 meters. In addition, oxygen saturation and heart rate, resting fatigue and dyspnea levels will be evaluated with pulse oximetry before and after testing. Modified Borg Dyspnea and Fatigue Scales will be used to determine resting dyspnea and fatigue levels.
Peak Expiratory Flow | 8 weeks
  Change of Expiratory Flow (PEF) from baseline to 8 weeks.
Forced Expiratory Volume in 1 second | 8 weeks
  Change of Forced Expiratory Volume in 1 second (FEV1) from baseline to 8 weeks.
Control of Asthma | 8 weeks
  Change of Asthma Control Test from baseline to 8 weeks. The Asthma Control Test is a 5-item questionnaire that enables the patient to assess his / her own level of exposure to asthma activities, frequency of day and night asthma symptoms, need for rescue medication, and disease control. Patients will be asked to answer the asthma control test, which includes scores associated with the answer to each question, and the total score will be 25 if complete control, 20-24 as partial control, and <19 as uncontrolled.
Dyspnoea | 8 weeks
  Change of Medical Research Council Scale results from baseline to 8 weeks. The Medical Research Council Scale (MRCS) is a five-item scale based on various physical activities that produce dyspnea. Here, patients are asked to mark the level of activity that causes dyspnea in themselves. On the scale, 0 describes the best 4 dyspnea and the worst.

SECONDARY OUTCOMES:
Lower Extremity Strength and Dynamic Balance | 8 weeks
  Change of 30 seconds sit and stand test results from baseline to 8 weeks.
Health Related Quality of Life | 8 weeks
  Change of Saint George Respiratory Questionnaire Results from baseline to 8 weeks.It is a self-answered questionnaire consisting of three categories, evaluating the symptoms, activities and effects of patients on daily life. It was developed in order to determine the severity of the disease as more comprehensive and sensitive. Symptoms examined; cough, sputum, wheezing and shortness of breath. Physical functions, housework and hobbies are questioned to determine activity status. The survey consists of 76 questions and is completed in 20 minutes. 0 indicates excellent health and 100 indicates worst health.
Activity of Daily Living | 8 weeks
  Change of London Chest Activity of Daily Living Scale results from baseline to 8 weeks. This questionnaire consisting of 15 items; personal care (4 items-dry, dress up upper body, wear shoes / socks, wash hair), housework (make 6 items-bed, change sheets, window / curtain wash, clean / remove dust, wash dishes, sweep), physical activity (2 items-stairs, leaning) and leisure (3 items-walking in the house, socially go out, talk) consists of four components. Each item is given a score ranging from 0 to 5. Higher scores indicate higher limitation. The scale can be evaluated as total score, component score and question score. The total score can reach up to 75.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Sena Manzak, PhD Student, Principal Investigator — Bezmialem Vakif University; Semiramis Özyılmaz, Assoc. Prof., Study Director — Bezmialem Vakif University
Locations (2):
- Turkey (Türkiye) (2):
  - Bezmialem Vakıf University, Istanbul, Eyüp
  - Bahçelievler Public Hospital, Istanbul